CLINICAL TRIAL: NCT01045499
Title: Laparoscopic Adjustable Gastric Banding (LAGB) as a Treatment for Morbid Obesity in Adolescents
Brief Title: LAGB as a Treatment for Morbid Obesity in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeffrey L Zitsman, MD (Other)
Responsible Party: Sponsor-Investigator, Jeffrey L Zitsman, MD, Professor of Surgery, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAB1759
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-03

CONDITIONS: Morbid Obesity; Obstructive Sleep Apnea Syndrome; Metabolic Syndrome; Insulin Resistance; Nonalcoholic Fatty Liver Disease
Keywords: adolescent obesity surgery; bariatric surgery; adjustable gastric banding
MeSH Terms: conditions — Obesity, Morbid; Sleep Apnea, Obstructive; Metabolic Syndrome; Insulin Resistance; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- laparoscopic gastric banding (Experimental): Adolescent patients who have undergone laparoscopic adjustable gastric banding. Weight, BMI, and co-morbidity data will be compared to patient's pre-operative values.
  Interventions: Device: Laparoscopic adjustable gastric banding (Allergan Lap Band)

INTERVENTIONS:
Device: Laparoscopic adjustable gastric banding (Allergan Lap Band) — Pre-op evaluation, surgical placement of a gastric band, and follow-up for a minimum of 5 years after surgery. Surgery is laparoscopic adjustable gastric band placement using a single brand of gastric band. Evaluations before and after surgery include but are not limited to history and physical examination, serum chemistry studies, imaging, sleep studies, and pulmonary function testing.
  Other Names: LAP-BAND®

SUMMARY:
Laparoscopic adjustable gastric banding (LAGB) has been used worldwide to help selected morbidly obese adults to lose weight. The FDA has approved LAGB only for patients 18 years or older. Our hypothesis that LAGB can be used to assist selected adolescents between 14 and 17 years lose weight and that the procedure can be performed safely in this age group. We are also evaluating the effects of weight loss after LAGB on known comorbid conditions such as sleep apnea syndrome and insulin resistance, and also on psychological health.

DETAILED DESCRIPTION:
Seventy to ninety-eight percent of obese children become obese adults. Comorbidities of obesity such as type II diabetes, fatty liver disease, hyperlipidemia, hypertension, asthma, sleep apnea, and depression are becoming increasing common in adolescents as more adolescents become obese. The only consistently durable and effective weight loss programs for the morbidly obese patients are those that include bariatric surgical procedures. The investigators believe that the best initial bariatric surgical option for adolescents is LAGB because of its low complication rates, adjustability, and reversibility. Obese adolescents ages 14-17 who meet criteria for entry will be enrolled to determine the degree of success of LAGB as measured by % excess weight loss, decreased % body fat, decreased body mass index (BMI), reduction in comorbid conditions, and metabolic parameters (including serum lipids and glucose tolerance) at intervals of 3 months, 6 months, 1 year, then annually for a total of 5 years postoperatively. Eligible patients will have been followed for 6 months by physicians in the Center for Adolescent Bariatric Surgery and: 1) will attended a minimum of 75% of visits and 2) will have failed to lose at least 20% of excess weight. Following evaluation by the team (which will include evaluations by a nutritionist, an endocrinologist, a psychologist/psychiatrist, a pediatric nurse practitioner, and a surgeon) a patient may be offered LAGB.

ELIGIBILITY:
Inclusion Criteria:

* Ages 13-17 upon entry
* BMI >40 or >35 with associated medical comorbidities (e.g., sleep apnea, hypertension

Exclusion Criteria:

* severe psychiatric illness
* eating disorder with purging
* previous weight loss surgery
* stated inability to comply with pre-op and post-op visits

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 137 (Actual)
Dates: Start 2005-09-13 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Zitsman, MD, Principal Investigator — Columbia University
Locations (1):
- Morgan Stanley Children's Hospital of NY Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sysko R, Devlin MJ, Hildebrandt TB, Brewer SK, Zitsman JL, Walsh BT. Psychological outcomes and predictors of initial weight loss outcomes among severely obese adolescents receiving laparoscopic adjustable gastric banding. J Clin Psychiatry. 2012 Oct;73(10):1351-7. doi: 10.4088/JCP.12m07690. PMID 23140654
- [Derived] Sysko R, Zakarin EB, Devlin MJ, Bush J, Walsh BT. A latent class analysis of psychiatric symptoms among 125 adolescents in a bariatric surgery program. Int J Pediatr Obes. 2011 Aug;6(3-4):289-97. doi: 10.3109/17477166.2010.545411. Epub 2011 Feb 8. PMID 21299450

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adolescents aged 13 to 18 years were enrolled in this study.
Pre-assignment Details: The age range for the enrolled adolescents at the time of surgery was 14-19 years of age since some aged from the time of consent to surgery.
Period: Overall Study
Arm/Group | Laparoscopic Gastric Banding
Started | 137
Completed | 127
Not Completed | 10

BASELINE CHARACTERISTICS:
Population: adolescents with morbid obesity 14-18yr
Groups:
- Adolescents With Morbid Obesity: At the time of enrollment, the adolescents with morbid obesity were aged 13-18 years of age and at the time of surgery, the adolescents were aged 14-19 years of age.
Arm/Group | Adolescents With Morbid Obesity
Number analyzed (Participants) | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.0 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 59
  More than one race | 4
  Unknown or Not Reported | 51
Family obesity [Count of Participants; unit: Participants]
  Mother | 34
  Father | 14
  Both | 31
  Yes (not identified) | 6
  Neither | 50
  Adopted (no information) | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Excess Weight Change (EWL)
Description: Weight change evaluated in terms of % excess weight loss (EWL).
Time Frame: Baseline and up to 5 years from start of study.
Population: Includes individuals with confirmed band status at 5 years after surgery.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Laparoscopic Gastric Banding
Number analyzed (Participants) | 127
percent change | -35.5 (39.4)

2. Secondary Outcome: Percentage of Excess BMI Change
Description: Change in Body mass index (BMI) in terms of excess BMI loss (EBMIL).
Time Frame: Baseline and up to 5 years from start of study.
Population: Includes individuals with confirmed band status at 5 years after surgery.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Laparoscopic Gastric Banding
Number analyzed (Participants) | 127
percent change | 36.6 (37.5)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded as perioperative if occurring less than or equal to 30 days following surgery and post-operative if greater than 30 days. Safety data was collected up to 5 years post-surgery.
Arm/Group | Laparoscopic Gastric Banding
All-Cause Mortality (participants affected / at risk) | 3/137
Serious Adverse Events (participants affected / at risk) | 63/137
Other Adverse Events (participants affected / at risk) | 137/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laparoscopic Gastric Banding (N=137)
Band removal due to dysphagia, reflux or heartburn (Surgical and medical procedures) | 3 (3)
Hiatal hernia repair (Surgical and medical procedures) | 1 (1)
Gastric Herniation (band slippage) (Surgical and medical procedures) | 10 (10)
Port site bleeding (Surgical and medical procedures) | 1 (1) — Resulted in surgery
Malpositioned band (Surgical and medical procedures) | 1 (1) — Resulted in surgery
Intestinal obstruction (Surgical and medical procedures) | 1 (1) — Resulted in surgery.
Port displacement (Surgical and medical procedures) | 11 (11) — Resulted in operative port repositioning.
Band removal (Surgical and medical procedures) | 33 (33)
Weight loss procedure (conversion) (Surgical and medical procedures) | 16 (16)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laparoscopic Gastric Banding (N=137)
Emesis (Gastrointestinal disorders) | 96 (266)
Abdominal pain (Gastrointestinal disorders) | 62 (114)
Port site pain (General disorders) | 46 (73)
GERD/Heartburn (Gastrointestinal disorders) | 44 (68)
Dysphagia/food stuck (Metabolism and nutrition disorders) | 40 (76)
Upper respiratory infection (URI) (Infections and infestations) | 32 (40)
Diarrhea (Gastrointestinal disorders) | 18 (25)
Headaches (General disorders) | 14 (16)
Sore throat (General disorders) | 14 (15)
Back pain (General disorders) | 12 (12)
Elevated CES-D Score (General disorders) | 12 (12)
Band slip/prolapse (Surgical and medical procedures) | 10 (14)
Port displacement/flip (Surgical and medical procedures) | 9 (10)
Dehydration (General disorders) | 8 (8)
Knee pain (General disorders) | 8 (11)
Esophagitis (Metabolism and nutrition disorders) | 8 (9)
Esophageal dilation (General disorders) | 7 (9)
Sinusitis (Infections and infestations) | 7 (8)
Fever (Infections and infestations) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes